CLINICAL TRIAL: NCT00849602
Title: The Effect of Chloroquine in the Treatment of Patients With Dengue
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Benedito Antonio Lopes da Fonseca, São Paulo University Medical School at Ribeirão Preto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BALF-01
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Placebo — Placebo bid for three days
  Arms: 1
Drug: Chloroquine — Chloroquine bid for three days
  Arms: 2

SUMMARY:
The objective of this study was to evaluate the effect of chloroquine in the treatment of patients with dengue.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of having dengue disease
* Patients were included in the study if they presented with fever and at least two other symptoms, such as:

  * headache
  * pain behind the eyes
  * muscle and bone or joint pains
  * nausea
  * vomiting
  * rash associated to dengue for less than 72 hours

Exclusion Criteria:

* Pregnant
* Younger than 18-years old
* Either cardiac or neurologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-05 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Duration of the disease | one week

SECONDARY OUTCOMES:
Intensity and days of fever and symptoms | one week

CONTACTS AND LOCATIONS:
Overall Officials: Benedito AL Fonseca, PhD, Principal Investigator — São Paulo University Medical School at Ribeirão Preto
Locations (1):
- São Paulo University Medical School at Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil